CLINICAL TRIAL: NCT00764517
Title: Phase II Study of Vorinostat (SAHA), Cladribine, and Rituximab (SCR) in Mantle Cell Lymphoma, Chronic Lymphocytic Leukemia, and Relapsed B Cell Non-Hodgkin Lymphoma
Brief Title: Vorinostat, Cladribine, and Rituximab in Treating Patients With Mantle Cell Lymphoma, Relapsed Chronic Lymphocytic Leukemia, or Relapsed B Cell Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Stephen Spurgeon, Associate Professor, OHSU Knight Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00004180; NCI-2011-03737 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 4180 (Other: OHSU IRB); HEM-08002-L (Other: OHSU Knight Cancer Insitute); CR00021415; IRB00004180 (Other: OHSU Knight Cancer Institute); P30CA069533 (NIH)
Record Dates: First submitted 2008-10-01; First posted 2008-10-02 (Estimated); Results first posted 2017-11-13 (Actual); Last update posted 2017-12-11 (Actual); Status verified 2017-10

CONDITIONS: Recurrent B-Cell Non-Hodgkin Lymphoma; Recurrent Chronic Lymphocytic Leukemia; Recurrent Indolent Adult Non-Hodgkin Lymphoma; Refractory B-Cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Cladribine; Rituximab; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Previously untreated (Experimental): Patients enrolled with untreated, newly diagnosed mantle cell lymphoma (MCL) or chronic lymphocytic leukemia (CLL) [Group I].
  Patients receive vorinostat PO on days 1-14, cladribine IV over 2 hours on days 1-5, and rituximab IV on day 3 (weekly for the first course). Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cladribine; Other: Laboratory Biomarker Analysis; Biological: Rituximab; Drug: Vorinostat
- Relapsed (Experimental): Patients with relapsed disease including indolent Non-Hodgkins Lymphoma (NHL), mantle cell lymphoma (MCL), or chronic lymphocytic leukemia (CLL) [Group II].
  Patients receive vorinostat PO on days 1-14, cladribine IV over 2 hours on days 1-5, and rituximab IV on day 3 (weekly for the first course). Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cladribine; Other: Laboratory Biomarker Analysis; Biological: Rituximab; Drug: Vorinostat

INTERVENTIONS:
Drug: Cladribine — Given IV
  Other Names: 2-CdA; 2CDA; CdA; Cladribina; Leustat; Leustatin; Leustatine; RWJ-26251
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Rituximab — Given IV
  Other Names: BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab Biosimilar BI 695500; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; RTXM83
Drug: Vorinostat — Given PO
  Other Names: L-001079038; SAHA; Suberanilohydroxamic Acid; Suberoylanilide Hydroxamic Acid; Zolinza

SUMMARY:
This phase II trial studies how well giving vorinostat, cladribine, and rituximab together works in treating patients with mantle cell lymphoma (MCL), chronic lymphocytic leukemia (CLL), or B cell non-Hodgkin's lymphoma (NHL) that has returned after a period of improvement. Vorinostat may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as cladribine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Monoclonal antibodies, such as rituximab, may block cancer growth in different ways by targeting certain cells. Giving vorinostat together with cladribine and rituximab may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine objective response rates of the SCR regimen (vorinostat, cladribine, and rituximab) in B-cell malignancies.

II. Determine the tolerability and toxicities of the SCR regimen.

SECONDARY OBJECTIVES:

I. Evaluate progression free survival in patients treated with SCR. II. Estimate event free survival for patients treated with SCR. III. Determine the contribution (if any) of deoxyribonucleic acid (DNA) methylation/histone deacetylation to disease progression and/or response to SCR combination chemotherapy.

IV. Perform scientific correlates to determine if SCR treatment a) is associated with global and gene specific changes in transcription of messenger ribonucleic acid (mRNA)s and micro ribonucleic acid (MiRNA)s b) is acting as an inhibitor of DNA methylation c) is activating or silencing specific genes or miRNAs.

OUTLINE:

Patients receive vorinostat orally (PO) on days 1-14, cladribine intravenously (IV) over 2 hours on days 1-5, and rituximab IV on day 3 (weekly for the first course). Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 2 years and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be able to provide informed consent according to institutional guidelines
* Patients must have: 1) MCL; or 2) relapsed or refractory cluster of differentiation (CD)20 positive B-cell indolent NHL; or 3) relapsed CLL
* Patients must have measurable disease/disease status requirements as follows:
* For CLL patients, symptomatic disease as defined by the International Workshop on Chronic Lymphocytic Leukemia (IWCLL) 2008 criteria that mandate treatment
* For B-cell NHL patients must have at least one of the following to be eligible:

  * Positron emission tomography (PET) avid or measurable disease by computed tomography (CT) scan defined as at least 1 lesion that measures > 2 cm in a single dimension
  * Significant bone marrow and/or peripheral blood involvement by NHL (i.e. leukemic phase) as determined by the investigator
  * Patients with Waldenström macroglobulinemia (WM) are exempt from this requirement if they have symptomatic hyperviscosity or clinically relevant cytopenias and elevated serum immunoglobulin M (IgM)
* Patients must have adequate bone marrow reserve as indicated by an absolute neutrophil count (ANC) > 1.500/mm^3 and platelet count > 150.000/mm^3 if no bone marrow involvement; however, if there is significant lymphoma/leukemia bone marrow infiltration, no pre-existing hematologic parameters must be met
* Patients must have a performance status of 0, 1, or 2 according to Eastern Cooperative Oncology Group
* Serum creatinine < 2.0 mg/dL or estimated glomerular filtration rate (GFR) > 60 mL/min
* Serum bilirubin =< 1.5 × upper limit of normal (ULN)
* Aspartate transaminase (AST)/alanine transaminase (ALT) =< 2.5 × ULN
* Alkaline phosphatase =< 2.5 × ULN
* Female patients of childbearing potential must have a negative serum pregnancy test within 2 weeks prior to enrollment
* Male and female patients must agree to use an effective contraceptive method during the study and for a minimum of 6 months after study treatment

Exclusion Criteria:

* Significant hypersensitivity to cladribine or vorinostat; hypersensitivity to rituximab infusion is not an exclusion criterion; however, appropriate changes to infusion schedules will be made based on current or prior reactions
* Current concomitant chemotherapy, radiation therapy, or immunotherapy other than as specified in the protocol
* Patients with a diagnosis of a relapsed/refractory aggressive cluster of differentiation antigen 20 (CD20)+ B-cell neoplasm defined as Burkitt's lymphoma or diffuse large B-cell lymphoma
* A diagnosis of acute lymphoplasmic leukemia, and lymphoblastic lymphoma
* Use of investigational agents or any anticancer therapy within 2 weeks before study entry with the exception of hydroxyurea and steroids; the patient must have recovered from all acute toxicities from any previous therapy
* Have any other severe concurrent disease, or have a history of serious organ dysfunction or disease involving the heart, kidney, liver, or other organ system that may place the patient at undue risk to undergo treatment
* Patients with a systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment)
* Pregnant or lactating patients
* Any significant concurrent disease, illness, or psychiatric disorder that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results
* Patients with acquired immunodeficiency syndrome (AIDS) or human immunodeficiency virus (HIV) associated complex are not eligible for treatment
* Patients with active hepatitis B or C are not eligible for the study
* Patients taking other histone deacetylases (HDAC) inhibitors; for example, patients taking valproic acid, there must be a 14 day washout period prior to enrollment in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2008-08; Primary Completion 2015-01 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Spurgeon, Principal Investigator — OHSU Knight Cancer Institute
Locations (2):
- United States (2):
  - OHSU Knight Cancer Institute, Portland, Oregon
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania

REFERENCES:
- [Derived] Spurgeon SE, Sharma K, Claxton DF, Ehmann C, Pu J, Shimko S, Stewart A, Subbiah N, Palmbach G, LeBlanc F, Latour E, Chen Y, Mori M, Hasanali Z, Epner EM. Phase 1-2 study of vorinostat (SAHA), cladribine and rituximab (SCR) in relapsed B-cell non-Hodgkin lymphoma and previously untreated mantle cell lymphoma. Br J Haematol. 2019 Sep;186(6):845-854. doi: 10.1111/bjh.16008. Epub 2019 Jun 9. PMID 31177537

RESULTS

PARTICIPANT FLOW:
Groups:
- Previously Untreated: Patients enrolled with untreated, newly diagnosed mantle cell lymphoma (MCL) or chronic lymphocytic leukemia (CLL) [Group I].
  Patients receive 400 mg vorinostat PO on days 1-14, 5 mg/m^2 cladribine IV over 2 hours on days 1-5, and 375 mg/m^2 rituximab IV on day 3 (weekly for the first course). Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
- Relapsed: Patients with relapsed disease including indolent Non-Hodgkins Lymphoma (NHL), mantle cell lymphoma (MCL), or chronic lymphocytic leukemia (CLL) [Group II].
  Patients receive 400 mg vorinostat PO on days 1-14, 5 mg/m^2 cladribine IV over 2 hours on days 1-5, and 375 mg/m^2 rituximab IV on day 3 (weekly for the first course). Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Previously Untreated | Relapsed
Started | 39 | 18
Completed | 24 | 4
Not Completed | 15 | 14
Not completed — Adverse Event | 9 | 3
Not completed — Death | 3 | 11
Not completed — Physician Decision | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Previously Untreated | Relapsed | Total
Number analyzed (Participants) | 39 | 18 | 57
Age, Continuous [Median (Full Range); unit: years] | 62 [35 to 87] | 60 [46 to 85] | 61.5 [35 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 34 | 15 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 37 | 18 | 55
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 37 | 18 | 55
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 39 | 18 | 57

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: ORR defined as the percentage of patients who achieved a complete response (CR) or a partial response (PR). Assessed per the revised Cheson criteria. Response definitions per revised International Working Group Response Criteria. 95% confidence interval will be provided. Definitions: Complete response (CR) = disappearance of all evidence of disease; Partial response (PR) = regression of measurable disease and no new sites.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Previously Untreated | Relapsed
Number analyzed (Participants) | 39 | 18
percentage of participants | 97 [87 to 100] | 39 [17 to 64]

2. Primary Outcome: Toxicities as Assessed Using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0
Description: Toxicity is determined percentage of patients that experienced an adverse event (AE) grade 3 or higher during the time frame, assessed using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Grade refers to the severity of the AE increasing from Grade 1 to 5. Generally, Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe or medically significant but not immediately life-threatening; Grade 4 = Life-threatening consequences; Grade 5 = Death related to AE.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Previously Untreated | Relapsed
Number analyzed (Participants) | 39 | 18
percentage of participants | 90 [76 to 97] | 83 [59 to 96]

3. Primary Outcome: Tolerability of Treatment
Description: Tolerability is determined to be the percentage of patients who completed the full duration of treatment (all 6 cycles) regardless of adverse event status. % tolerability shows the rate of patients that tolerated the treatment for the full duration.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Previously Untreated | Relapsed
Number analyzed (Participants) | 39 | 18
percentage of participants | 62 [45 to 77] | 22 [6 to 48]

4. Secondary Outcome: Progression-free Survival
Description: Time from treatment start until disease progression or death.
  Estimated using the Kaplan-Meier method. A logrank test will be used to compare progression-free survival between Group I and Group II. A p-value less that 0.05 will be considered statistically significant.
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Previously Untreated | Relapsed
Number analyzed (Participants) | 39 | 18
Months | NA [25 to NA] — Median survival not reached. Upper confidence limit is inestimable. | 19.5 [2 to 33]
Statistical Analysis 1: Comparison: Previously Untreated vs Relapsed; Test type: Other; p = 0.002, Log Rank; Hazard Ratio (HR) = 0.33, 95% CI 2-sided [0.16 to 0.69]

5. Secondary Outcome: Event-free Survival
Description: Time from treatment start until disease progression, death, or discontinuation of treatment for adverse event (toxicity)
  Estimated using the Kaplan-Meier method. A logrank test will be used to compare progression-free survival between Group I and Group II. A p-value less that 0.05 will be considered statistically significant.
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Previously Untreated | Relapsed
Number analyzed (Participants) | 39 | 18
Months | 39.0 [25 to NA] — Upper confidence limit is inestimatable | 19.5 [2.0 to 34.0]
Statistical Analysis 1: Comparison: Previously Untreated vs Relapsed; Test type: Other; p = 0.011, Log Rank; Hazard Ratio (HR) = 0.42, 95% CI 2-sided [0.21 to 0.84]

6. Secondary Outcome: Contribution (if Any) of DNA Methylation/Histone Deacetylation
Description: Determine the contribution (if any) of DNA methylation/histone deacetylation to disease progression and/or response to SCR combination chemotherapy.
  Outcome not evaluated due to technical challenges collecting the data, and lack of budget and personnel to complete the analysis.
Time Frame: Up to 2 years
Population: Data not collected and the outcome will never be analyzed.
Arm/Group | Previously Untreated | Relapsed
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Scientific Correlates
Description: Perform scientific correlates to determine if SCR treatment a) is associated with global and gene specific changes in transcription of mRNAs and MiRNAs b) is acting as an inhibitor of DNA methylation c) is activating or silencing specific genes or miRNAs.
  Outcome not evaluated due to technical challenges collecting the data, and lack of budget and personnel to complete the analysis.
Time Frame: Baseline
Population: Data not collected and the outcome will never be analyzed.
Arm/Group | Previously Untreated | Relapsed
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 25 weeks (6 cycles X 28 days + 1 week after last cycle. Toxicities and adverse experiences will be assessed at each visit using the NCI Common Terminology Criteria for Adverse Events v4.0. Adverse events evaluated and recorded using the NCI CTCAE, Version 4.0 for 1 week after last cycle.
Description: For reporting purposes here, Grade 4 will be considered to be serious adverse event (SAE).
  Events assessed at each visit during the study (every other week for Cycle 1, then monthly for Cycles 2 to 6)
Arm/Group | Previously Untreated | Relapsed
All-Cause Mortality (participants affected / at risk) | 8/39 | 13/18
Serious Adverse Events (participants affected / at risk) | 18/39 | 9/18
Other Adverse Events (participants affected / at risk) | 28/39 | 14/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Previously Untreated (N=39) | Relapsed (N=18)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Cardiac troponin I increased (Investigations) | 1 (1) | 0 (0)
Death NOS (General disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
INR increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 9 (10) | 4 (4)
Platelet count decreased (Investigations) | 4 (4) | 4 (4)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Previously Untreated (N=39) | Relapsed (N=18)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Aortic valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac troponin I increased (Investigations) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 5 (5) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 9 (11) | 5 (5)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
heart failure (Cardiac disorders) | 1 (1) | 0 (0)
Hemoglobin decreased (Investigations) | 1 (1) | 1 (1)
Hemoglobin increased (Investigations) | 0 (0) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (3) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Infection: pulmonary (lung) (Infections and infestations) | 0 (0) | 1 (1)
Infusion related reaction (General disorders) | 1 (1) | 0 (0)
INR increased (Investigations) | 1 (1) | 1 (1)
Neutrophil count decreased (Investigations) | 7 (8) | 5 (6)
Pain (General disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 14 (15) | 5 (5)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 2 (2) | 0 (0)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Weight loss (Investigations) | 2 (2) | 1 (1)

LIMITATIONS AND CAVEATS:
Secondary objectives and outcomes not evaluated due to technical challenges collecting the data, and lack of budget and personnel to complete the analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No